CLINICAL TRIAL: NCT00004097
Title: A Phase I Study of Concomitant Chemoradiotherapy With Gemcitabine, Paclitaxel, and 5-FU for Patients With Advanced and/or Recurrent Cancer of the Head and Neck
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Advanced and/or Recurrent Head and Neck Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: NU C97N2; NU-C97N2; NCI-G99-1590
Record Dates: First submitted 1999-12-10; First posted 2004-03-31 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-10

CONDITIONS: Head and Neck Cancer
Keywords: stage III nasopharyngeal cancer; stage IV nasopharyngeal cancer; recurrent nasopharyngeal cancer; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; stage III lip and oral cavity cancer; stage IV lip and oral cavity cancer; recurrent lip and oral cavity cancer; stage III hypopharyngeal cancer; stage IV hypopharyngeal cancer; recurrent hypopharyngeal cancer; stage III laryngeal cancer; stage IV laryngeal cancer; recurrent laryngeal cancer; stage III paranasal sinus and nasal cavity cancer; stage IV paranasal sinus and nasal cavity cancer; recurrent paranasal sinus and nasal cavity cancer; stage III oropharyngeal cancer; stage IV oropharyngeal cancer; recurrent oropharyngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Nasopharyngeal Neoplasms; Mouth Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Oropharyngeal Neoplasms | interventions — Fluorouracil; Gemcitabine; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating patients who have advanced and/or recurrent head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of gemcitabine when administered with paclitaxel and fluorouracil with concurrent hyperfractionated radiotherapy in patients with advanced and/or recurrent head and neck cancer. II. Determine the MTD and DLT of gemcitabine as a single agent with radiotherapy in these patients. III. Determine the efficacy of concurrent chemoradiotherapy in terms of time to progression, pattern of failure, and overall survival in patients with measurable disease. IV. Determine gemcitabine and fluorouracil pharmacokinetics in these patients.

OUTLINE: This is a dose escalation study of gemcitabine, conducted in two phases. Phase A: Patients receive fluorouracil IV continuously on days 1-5, paclitaxel IV over 1 hour on day 2, and radiotherapy administered twice daily on days 1-5. This regimen is repeated every 2 weeks for 2 courses, then gemcitabine IV over 30 minutes is added on day 2 after paclitaxel. This regimen is administered every 2 weeks for 3 courses. Patients with responsive disease may continue chemotherapy (without radiotherapy) for 2 courses beyond maximum response. Cohorts of 3-6 patients receive escalating doses of gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 3 of 6 patients experience dose-limiting toxicity. Phase B: After the MTD of gemcitabine is determined in phase A, further dose escalation of gemcitabine may be performed with concurrent radiotherapy (without fluorouracil or paclitaxel). The MTD is determined as in phase A. Patients are followed monthly for 1 year and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 30-40 patients will be accrued for this study within approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven head and neck cancer requiring regional radiotherapy Locoregional, recurrent disease after primary therapy with surgery, radiation, or both OR Stage IV, no prior therapy, and not amenable to conventional therapy with curative intent Metastatic disease allowed if predominant site and associated symptoms require local treatment in the head and neck region

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC greater than 3,000/mm3 Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception No significant infection No other severe medical illness

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Recovered from any prior chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Recovered from any prior radiotherapy Surgery: See Disease Characteristics Recovered from any prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Argiris, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (2):
- United States (2):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois